CLINICAL TRIAL: NCT04135391
Title: Effects of Aerobic Interval Exercise Training on Cardiac Fibroblasts and Brain Cells in Stroke Patients
Brief Title: Aerobic Trainings on Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201600576A3
Record Dates: First submitted 2019-10-20; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-07

CONDITIONS: Stroke, Cardiovascular
Keywords: Stroke; Oxygen consumption; BDNF; Dendrites
MeSH Terms: conditions — Myocardial Infarction; Stroke

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial was performed in stroke patients adequate for exercise trainings. Different exercise regimens were prescribed and was blind to the assessors. The study was conducted from August 2016 to June 2018. Participants were randomly allocated to the moderate-intensity continuous training (MICT) or high-intensity interval training (HIIT) groups using a computer-generated, concealed allocation schedule. All included stroke patients received traditional rehabilitation programs, including balance, range of motion, or therapeutic exercise, and additional in-hospital supervised 30 min of MICT or HIIT for 36 times. Data were collected by a blinded assessor prior to randomization after completing the exercise trainings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pre- and Post- exercise training effects (Experimental): All recruited subjects received aerobic exercise training (HIIT or MICT). VO2peak, cardiac output (CO), bilateral frontal cortex blood volume (∆[THb]), oxyhemoglobin (∆[O2Hb]) and deoxyhemoglobin (∆[HHb]), ventilation efficiency, serum brain-derived neurotrophic factor (BDNF) levels, cognitive and life quality questionnaire, percentage of neuroblastic cell bearing neurites (% neurites), and cell fluorescent staining were examined before and after interventions.
  Interventions: Behavioral: Aerobic exercise training

INTERVENTIONS:
Behavioral: Aerobic exercise training — All recruited subjects underwent 36 times of moderate-intensity continuous training (MICT) at 60% of peak oxygen consumption (VO2peak) for 30 mins, and 10or had high-intensity interval training (HIIT) at alternative 80% and 40% VO2peak with the same training times and duration.

SUMMARY:
Effects of different exercise strategies on stroke patients remain unclear. Randomized controlled trial with concealed allocation has been performed from August 1, 2016 to June 30, 2018. We traced back 23 stroke patients, recruited during the above period, aged about 55 years with stroke duration > 24 months . Intervention: 13 of them underwent 36 times of moderate-intensity continuous training (MICT) at 60% of peak oxygen consumption (VO2peak) for 30 mins, and 10 had high-intensity interval training (HIIT) at alternative 80% and 40% VO2peak with the same training times and duration. Outcome measures: VO2peak, cardiac output (CO), bilateral frontal cortex blood volume (∆[THb]), oxyhemoglobin (∆[O2Hb]) and deoxyhemoglobin (∆[HHb]), ventilation efficiency, serum brain-derived neurotrophic factor (BDNF) levels, cognitive and life quality questionnaire, percentage of neuroblastic cell bearing neurites (% neurites), and cell fluorescent staining were examined before and after interventions.

DETAILED DESCRIPTION:
Design The Institutional Review Board of a tertiary care hospital approved the study (IRB No. 201600576A3). A randomized controlled trial was performed in stroke patients with different exercise regimens and was blind to the assessors. The study was conducted from August 2016 to June 2018. Participants were randomly allocated to the MICT or HIIT groups using a computer-generated, concealed allocation schedule. All included stroke patients received traditional rehabilitation programs, including balance, range of motion, or therapeutic exercise, and additional in-hospital supervised 30 min of MICT or HIIT for 36 times. Data were collected by a blinded assessor prior to randomization after completing the exercise trainings.

Participants Stroke patients, diagnosed by the neurologist, were surveyed. The inclusion criteria were listed as follows: (I) ≥ 20 years old; (II) stroke events with stable clinical status ≥ 3 months; (III) mini-mental state examination (MMSE)> 24; (IV) no acute coronary syndrome. Those who had unstable angina, systolic blood pressure> 200 mmHg or diastolic blood pressure> 110 mm Hg, symptomatic orthostatic hypotension, severe aortic stenosis (peak systolic pressure gradient> 50 mmHg, or an aortic valve opening area< 0.75 cm2), inflammatory disease within recent 3 months, uncontrolled cardiac dysrhythmias, uncompensated HF, third degree atrioventricular block, pericarditis or myocarditis within recent 3 months, embolic disease within recent 3 months, ST segment displacement≥ 2 mm at rest, and uncontrolled diabetes (blood glucose≥ 300 mg/dL or ≥ 250 mg/dL with ketone bodies) were not candidates of the study.

Stroke patients had absolute contraindications for cardiopulmonary exercise test (CPET) and aerobic activities, suggested by the American College of Sports Medicine (ACSM), were also excluded in the study. Afterwards, eligible participants were randomly assigned to the MICT and HIIT groups. Baseline demographic characteristics were also recorded. All subjects provided informed consent after the experimental procedures were explained.

Cardiopulmonary exercise test (CPET) Participants underwent an incremental exercise test on a bicycle ergometer (Ergoselect 150P, ergoline GmbH, Bitz, Germany) and the examination was performed at a work-rate of 10 W/min with continuous monitoring heart rate, brachial blood pressure, and arterial oxygen saturation, until the stop conditions described previously. Oxygen consumption (VO2) was measured by a cardiopulmonary measurement device (MasterScreen CPX, CareFusion Corp., Hoechberg, Germany). The VO2peak, minute ventilation (VE), and carbon dioxide production (VCO2) were defined as the guideline for exercise testing suggested by the ACSM. VE and VCO2 responses, acquired from the initiation of exercise to the peak values, were used to calculate the VE-VCO2 slope using the least-square linear regression. The O2 uptake efﬁciency slope (OUES), an estimation of the O2 consumption efficiency during exercise, was derived from the slope of a natural logarithm plot of VE vs. VO2.

Cardiac hemodynamic measurements Noninvasive continuous cardiac output monitoring system (NICOM, Cheetah Medical, Wilmington, Delaware) was used to evaluate cardiac hemodynamic response to exercise, which analyzes the phase shift (ΔΦ) created by alternating electrical current across the chest of the subject as described in our previous study.

Cerebral hemodynamic measurements Two pairs of near infra-red spectroscopy (NIRS) probes (Oxymon, Artinis, The Netherland) were attached to bilateral frontal areas of each included subject during CPET. The Beer-Lambert law was applied to measure light absorption across each pair of NIRS detectors reflecting changes of oxyhemoglobin ([O2Hb]) and deoxyhemoglobin ([HHb]) in the frontal cortex during exercise. Total Hb amount ([THb]) was calculated as the sum of [O2Hb] and [HHb], and was used as an index of change in blood volume in the frontal cortex. Differences of the tissue oxygenation (Δ[O2Hb] and Δ[HHb]) and regional blood flow (Δ[THb]) between involved and uninvolved frontal cortices (involved-uninvolved) were used to estimate effects of different exercise regimens on brain tissue oxygenation and regional blood flow.

Health-related QoL QoL was measured by the Short Form-36 Health Survey questionnaire (SF-36), and mini-mental status examination (MMSE) was used to assess QoL and cognitive functions of the participants.

Exercise training protocols The included subjects underwent 36 times of supervised hospital-based training (2-3 session/week) on a bicycle ergometer (Ergoselect 150P, Germany) as our previous protocol.15 The training comprised a warm-up at 30% of VO2peak for 3 min, followed by a MICT (60% of VO2peak) or HIIT (five 3-min intervals at 80% of VO2peak and each interval separated by 3-min exercise at 40% of VO2peak) for 30 min, and then a cool-down at 30% of VO2peak for 3 min. The training was terminated when the subject had symptoms/signs suggested by the ACSM guideline.

Serum preparation An amount of 20 ml fresh blood was collected from all our subjects before and after exercise training. Samples were centrifuged at 2500 rpm for 5 min at room temperature, and the upper serum was preserved for cell culture and measurement of serum BDNF levels.

Measurement of serum BDNF BDNF levels were assessed before and after aerobic exercise trainings. Prepared serum of 100 µL was added in each well coated with the human BDNF capture antibody in a solid-phase sandwich, two-site enzyme linked immunoassay (ELISA) kit (BioVision Inc., Milpitas, CA). The BDNF level was then determined by the microplate reader (SpectraMax M3, Molecular Devices LLC, San Jose, CA).

Cell culture and neurite growth assay Rat neuroblastic cells (PC-12 cell line) were grown in Dulbecco's modified Eagle's medium (DMEM) supplemented with 7.5% patient serum (before and after exercise training), 7.5% horse serum (HS), 100 units/ml penicillin, and 100 mg/L streptomycin.

A total of 100000 cells were plated overnight on 35-mm dishes coated with poly- DL-lysine. After serum starvation in DMEM containing 2% HS for 12-18 h, cells were treated with 50 ng/ml NGF for the indicated time. Morphological changes were observed using the Leica TCS SP8 confocal microscopy 7 days after cultured with patient sera before and after exercise training. Percentage of cells with neurites of at least one cell body diameter in length was determined in five independent fields of every plate.

Fluorescent stains Cells (100000) were inoculated in each well of the eight-chamber slide (Millicell EZ slide, Millipore Corp., Billerica, MA) and were incubated at the pre- and post-MICT or HIIT sera for 12h. Vivid staining of Mitotracker (Invitrogen corp., Carlsbad, CA) was used to observe mitochondria in neuroblastic cells treated with sera from the above different status. The cells were stained with primary rabbit monoclonal anti-⍺-tubulin antibodies (Cell Signaling Technology Inc., Boston, MA). Fluorescein isothiocyanate-conjugated AffiniPure Goat anti-rabbit IgG (Jackson ImmunoResearch Laboratories, West Grove, PA) was used as the secondary antibody. Nuclei were counterstained with mounting medium (Vector Laboratories Inc., Burlingame, CA) containing 40,6-diamidino-2-phenylindole. The stained cells were examined with a confocal microscopic examination (Leica TCS SP8, Leica Microsystems Inc., Buffalo Grove, IL).

Statistical analysis Chi-square test was conducted to compare differences of non-parametric parameters between the two groups. Mann-Whitney U test was used to assess differences of age, stroke duration, body mass index (BMI), changes of exercise capacity, changes of brain oxygenation as well as regional blood volume, changes of BDNF levels, and changes of cell behaviors between the two groups. Differences of within group changes in numerical data was assessed by Wilcoxon matched-pair signed-rank test. Relationships between changes of measured clinical parameters after the exercise training and clinical information were analyzed by Pearson correlation. A p value < 0.05 was considered as statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients, diagnosed by the neurologist, with stable clinical status for greater than 3 months after conservative treatment or intervention were enrolled in the study.
* Mini-mental state examination (MMSE)> 24
* No acute coronary syndrome

Exclusion Criteria:

* Unstable angina
* Systolic blood pressure> 200 mmHg or diastolic blood pressure> 110 mm Hg
* Symptomatic orthostatic hypotension
* Severe aortic stenosis (peak systolic pressure gradient> 50 mmHg, or an aortic valve opening area< 0.75 cm2)
* Inflammatory disease within recent 3 months
* Uncontrolled cardiac dysrhythmias
* Uncompensated heart failure
* Pericarditis or myocarditis within recent 3 months
* Embolic disease within recent 3 months
* ST segment displacement≥ 2 mm at rest
* Uncontrolled diabetes (blood glucose≥ 300 mg/dL or ≥ 250 mg/dL with ketone bodies).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Peak cardiac output (CO) | 3-4 months (for 36 times of exercise training)
  Peak CO in millimeter per minute measured by non-invasive cardiac output measurement during exercise test before and after exercise training.
Peak exercise oxygen consumption (VO2peak) | 3-4 months (for 36 times of exercise training)
  VO2peak in ml/min/kg measured by cardiopulmonary function test before and after exercise training.
Oxygen uptake efficiency slope (OUES) | 3-4 months (for 36 times of exercise training)
  OUES in liter per minute/log(Liter per minute) derived from oxygen consumptions along time during exercise test before and after exercise training.
Ventilation/VCO2 ratio (Ve-VCO2) | 3-4 months (for 36 times of exercise training)
  Ve-VCO2, a number, derived from exhaled CO2 (ml/min/kg) versus ventilation (ml/min/kg) graph along time during exercise test before and after exercise training.
Differences of the brain tissue oxyhemoglobin (∆[O2Hb]) | 3-4 months (for 36 times of exercise training)
  Differences oxyhemoglobin between involved and uninvolved frontal cortices in μM measured by two pairs of near infra-red spectroscopy (NIRS) probes before and after exercise training.
Differences of the brain tissue deoxygenation (∆[HHb]) | 3-4 months (for 36 times of exercise training)
  Differences deoxyhemoglobin between involved and uninvolved frontal cortices in μM measured by two pairs of near infra-red spectroscopy (NIRS) probes before and after exercise training.
Differences of regional blood volume (∆[THb]) | 3-4 months (for 36 times of exercise training)
  Differences regional blood volume between involved and uninvolved frontal cortices in μM measured by two pairs of near infra-red spectroscopy (NIRS) probes before and after exercise training.
Physical component score (PCS) | 3-4 months (for 36 times of exercise training)
  Physical role function obtained from short form 36 questionnaire (SF-36) before and after exercise training. The SF-36 consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Mental component score (MCS) | 3-4 months (for 36 times of exercise training)
  Mental health score obtained from short form 36 questionnaire (SF-36) before and after exercise training. The SF-36 consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Mini-mental status examination (MMSE) | 3-4 months (for 36 times of exercise training)
  a 30-point questionnaire that is used extensively to measure cognitive impairment before and after exercise training.
Brain-derived neurotrophic factor (BDNF) | 3-4 months (for 36 times of exercise training)
  The human BDNF (ng/mL), essential in maintaining neurogenesis and synaptic plasticity, capture antibody in a solid-phase sandwich, two-site enzyme linked immunoassay (ELISA) kit. The BDNF level was then determined by the microplate reader before and after exercise training.
Percentage of cell bearing neurites | 3-4 months (for 36 times of exercise training)
  A total of 100000 cells were plated overnight on 35-mm dishes coated with poly- DL-lysine. After serum starvation in DMEM containing 2% HS for 12-18 h, cells were treated with 50 ng/ml NGF for the indicated time. Morphological changes were observed using the Leica TCS SP8 confocal microscopy 7 days after cultured with patient sera before and after exercise training. Percentage of cells with neurites of at least one cell body diameter in length was determined in five independent fields of every plate.
Neuron images | 3-4 months (for 36 times of exercise training)
  Cells (100000) were inoculated in each well of the eight-chamber slide (Millicell EZ slide, Millipore Corp., Billerica, MA) and were incubated at the pre- and post-MICT or HIIT sera for 12h. Vivid staining of Mitotracker (Invitrogen corp., Carlsbad, CA) was used to observe mitochondria in neuroblastic cells treated with sera from the above different status. The cells were stained with primary rabbit monoclonal anti-⍺-tubulin antibodies (Cell Signaling Technology Inc., Boston, MA). Fluorescein isothiocyanate-conjugated AffiniPure Goat anti-rabbit IgG (Jackson ImmunoResearch Laboratories, West Grove, PA) was used as the secondary antibody. Nuclei were counterstained with mounting medium (Vector Laboratories Inc., Burlingame, CA) containing 40,6-diamidino-2-phenylindole. The stained cells were examined with a confocal microscopic examination (Leica TCS SP8, Leica Microsystems Inc., Buffalo Grove, IL).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu CC, Fu TC, Huang SC, Chen CP, Wang JS. Increased serum brain-derived neurotrophic factor with high-intensity interval training in stroke patients: A randomized controlled trial. Ann Phys Rehabil Med. 2021 Jul;64(4):101385. doi: 10.1016/j.rehab.2020.03.010. Epub 2020 May 11. PMID 32344098